CLINICAL TRIAL: NCT01026129
Title: Efficacy of a Bolus Dose of Remifentanil Compared to a Bolus Dose of Intravenous lidocaïne on the Incidence of Coughing During Emergence of Anesthesia.
Brief Title: Efficacy of Remifentanil Compared to Lidocaine on the Incidence of Coughing During Emergence of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: François Girard, MD FRCPC, Centre de recherche du CHUM (CRCHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FG 2010-002
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Cough; Anesthesia; Extubation
MeSH Terms: conditions — Cough | interventions — Remifentanil; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Remifentanil 0.25 mcg/kg (Experimental): Administration of a bolus dose of remifentanil 0.25 mcg/kg before emergence of a desflurane-based anesthesia.
  Interventions: Drug: Remifentanil
- Remifentanil 0.5 mcg/kg (Experimental): Administration of a bolus dose of remifentanil 0.5 mcg/kg before emergence of a desflurane-based anesthesia.
  Interventions: Drug: Remifentanil
- Lidocaine (Active Comparator): Bolus dose of intravenous remifentanil 1mg/kg given once before emergence of general anesthesia.
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: Remifentanil — Bolus dose of intravenous remifentanil 0,25 mcg/kg given once before emergence of general anesthesia.
  Arms: Remifentanil 0.25 mcg/kg
Drug: Remifentanil — Bolus dose of intravenous remifentanil 0.5 mck/kg given once before emergence of general anesthesia.
  Arms: Remifentanil 0.5 mcg/kg
Drug: lidocaine — Bolus dose of intravenous remifentanil 0.5 mck/kg given once before emergence of general anesthesia.
  Arms: Lidocaine

SUMMARY:
This study is designed to compare the effects of a bolus dose of remifentanil to a bolus dose of lidocaine given prior to the emergence of anesthesia:

* on the incidence of perioperative coughing
* on the time needed for the emergence of a desflurane-based anesthesia
* on the incidence of sore throat after extubation.

Our hypothesis is that the use of a remifentanil bolus dose given prior to emergence of a desflurane-based anesthesia will reduce the incidence of perioperative coughing from 70% to 35% compared to lidocaine.

DETAILED DESCRIPTION:
Emergence is an important period of general anesthesia during which several problems can occur. Coughing, hypertension, tachycardia and agitation have been observed during emergence of general anesthesia.

Most patients will cough during emergence. Different techniques and drugs have been studied to reduce coughing during emergence. Among others, the role of lidocaine given intravenously, topically , or intra-cuff has been studied.

There is some evidence supporting the administration of intravenous opioids prior to emergence of general anesthesia to reduce perioperative coughing, agitation and haemodynamic stimulation. However, depending on the type of opioids given, this may delay the emergence from anesthesia. The effect of a remifentanil infusion given in combination with isoflurane as the volatile agent has been shown to reduce the incidence of perioperative coughing without delaying the emergence of anesthesia. The effect of a small bolus of remifentanil given prior to emergence to prevent perioperative coughing has yet to be studied.

Desflurane is a newer volatile agent allowing early recovery from anesthesia. This agent has led to earlier discharge and more rapid resumption of normal activities after surgery. However, an incidence of coughing around 70% has been reported after a desflurane-based anesthesia.

This study will compare the effects of remifentanil (bolus dose of 0.25 mcg/kg or 0.5 mcg/kg) to lidocaine (bolus dose of 1mg/kg) when given prior to emergence to prevent perioperative coughing after a desflurane-based anesthesia.

Methods:

* Induction of general anesthesia: 1.5-3 mg/kg propofol and 1-3 mcg/kg fentanyl. Neuromuscular relaxation at the discretion of the attending anesthesiologist.
* Tracheal intubation using direct laryngoscopy.
* Maintenance of general anesthesia: desflurane between 0.7 and 1.0 MAC, fentanyl 1 mcg/kg. Neuromuscular relaxation will be carried out at the discretion of the attending anesthesiologist.
* No opioids should be given during the last 30 minutes of surgery.
* Reversal of neuromuscular blockade is mandatory at the end of surgery.
* At the end of surgery : discontinuation of desflurane.
* Administration of the study drug: (bolus dose of remifentanil 0.25 mcg/kg, remifentanil 0.5 mcg/kg or lidocaine 1 mg/kg).
* When the expired fraction of desflurane reaches 0.2 MAC, the patient will be asked to open his eyes every 30 seconds.
* After eyes opening, ventilator will be stopped and the extubation performed.
* Number of coughing episodes and their importance will be rated on a scale from 0 to 3 by a blinded observer during emergence and the first ten minutes after extubation.
* Time elapsed between the administration of the bolus dose of the study drug to extubation will be recorded.
* The presence of sore throat will be assessed one hour after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* ASA physical status 1-3
* Patients undergoing elective surgery under general anesthesia requiring endotracheal intubation (excluding head and neck surgery)

Exclusion Criteria:

* Current use of ACE inhibitor
* Chronic cough
* Asthma or severe COPD
* Pulmonary tract infection
* Anticipated difficult intubation
* Current use of opioids
* Current use of cough medicine
* Contraindication to remifentanil or lidocaine
* Pregnancy
* Symptomatic cardiac, renal or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing during emergence and the first ten minutes after extubation. | From emergence until 10 minutes after extubation

SECONDARY OUTCOMES:
Time elapsed between the bolus dose of remifentanil or lidocaine and extubation. | From the administration of the study drug until extubation.
Incidence of sore throat one hour after extubation. | Assessed one hour after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada